CLINICAL TRIAL: NCT03366259
Title: Does the Administration of Prostaglandins Before Cesarean Section Reduce the Amount of Blood Loss ?
Brief Title: Prostaglandins Before Caserean Section
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, sarah mohamed hassan, lecturer of obstetrics and gynecology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4122017
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Intrapartum Hemorrhage
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Misoprostol group) (Active Comparator): 200 mcg rectal Misoprostol administration before cesarean section
  Interventions: Drug: Misoprostol 200Mcg Tab; Procedure: elective cesarean section
- Group B (control group) (Placebo Comparator): No prostaglandins administration before cesarean section
  Interventions: Procedure: elective cesarean section

INTERVENTIONS:
Drug: Misoprostol 200Mcg Tab — administration of 200 Mcg of misoprotol rectal
  Arms: Group A (Misoprostol group)
Procedure: elective cesarean section — elective cesarean section for full term patients

SUMMARY:
The aim of our study is to assess the value of administration of prostaglandins before cesarean section to reduce the amount of blood loss

DETAILED DESCRIPTION:
160 full term pregnant patients candidate for elective cesarean section were randomly allocated into 2 groups ,80 patients will receive 200mcg of rectal prostaglandins before cesarean section and 80 patients are used as control receiving placebo

ELIGIBILITY:
Inclusion Criteria:pregnant patients full term elective cesarean section

-

Exclusion Criteria:

* medical disorder with pregnancy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
amount of intraoperative blood loss | during cesarean section
  number of soaked towels
postpartum hemorrhage | 24 hour after cesarean section
  blood loss after cesarean section

SECONDARY OUTCOMES:
fetal condition | 5 minutes after cesarean section
  apgar score

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainiy Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No